CLINICAL TRIAL: NCT00494767
Title: An Exploratory Study to Evaluate Weight Loss, Body Composition Changes, Food Intake and Urine Glucose Excretion in Healthy Obese Subjects Over 8 Weeks of Dosing With GSK189075, GW869682 Versus Placebo
Brief Title: Investigation Of Weight Loss And Body Composition Changes After Dosing With Either Placebo Or One Of Two Active Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: KGW108201
Record Dates: First submitted 2006-10-31; First posted 2007-07-02 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: body composition; obesity; 4C model; hunger; weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GW869682 1000 mg thrice daily (TID) (Experimental): Subjects will be randomized to receive GW869682 1000 mg TID
  Interventions: Drug: GW869682; Drug: GSK189075; Drug: GSK189075-Placebo; Drug: GW869682-Placebo
- GSK189075 250 mg TID (Experimental): Subjects will be randomized to receive GSK189075 250 mg TID
  Interventions: Drug: GW869682; Drug: GSK189075; Drug: GSK189075-Placebo; Drug: GW869682-Placebo
- GW869682-Placebo TID (Placebo Comparator): Subjects will be randomized to receive Placebo matching GW869682 for TID
  Interventions: Drug: GW869682; Drug: GSK189075; Drug: GSK189075-Placebo; Drug: GW869682-Placebo
- GSK189075-Placebo TID (Placebo Comparator): Subjects will be randomized to receive Placebo matching GSK189075 for TID
  Interventions: Drug: GW869682; Drug: GSK189075; Drug: GSK189075-Placebo; Drug: GW869682-Placebo

INTERVENTIONS:
Drug: GW869682 — GW869682 tablet with a dose strength of 250 mg will be available for subjects
Drug: GSK189075 — GSK189075 tablet with a dose strength of 250 mg will be available for subjects
  Other Names: GW869682
Drug: GSK189075-Placebo — Placebo tablets to match GSK189075 250 mg will be available for subjects
Drug: GW869682-Placebo — Placebo tablets to match GW869682 250 mg will be available for subjects

SUMMARY:
The drugs GSK189075 and GW869682 result in increased caloric losses. This study is investigating how if taken over 8 weeks that affects weight loss, food intake and the composition of the body. The body composition (fat,water, lean mass) is determined using a new investigational MR technology.

ELIGIBILITY:
Inclusion criteria:

* BMI of 30 - 40kg/m
* Females may be included if they are surgically sterile or post-menopausal

Exclusion criteria:

* Change in body weight >4% in the last 3 months
* History of eating disorders
* had bariatric surgical intervention for obesity
* have type I or II diabetes
* Thyroid disorder not under control
* Renal or hepatobiliary disease
* Excessive alcohol consumption
* Use of drugs of abuse
* donated of blood in the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09-29 (Actual); Primary Completion 2007-06-07 (Actual); Study Completion 2007-06-07 (Actual)

PRIMARY OUTCOMES:
Body fat and fat-free mass as determined by a new investigational MR technique compared to 4C Model methodologies. | Measurements at week 8 will be compared to measurements from Day -1

SECONDARY OUTCOMES:
Safety (caloric losses body weight, body composition, weight and hip circumference.) | throughout study (Days 1-56)
Leptin levels in serum | at several points during study
Drug levels in blood over time (Day 42 PK parameters are AUC, Cmax, tmax) | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study KGW108201 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/KGW108201?search=study&search_terms=KGW108201#rs